CLINICAL TRIAL: NCT04013685
Title: A Phase Ib Trial of Patients With Advanced Hematologic Malignancies Undergoing Allogeneic Hematopoietic Cell Transplantation With Either Orca-T, a T-cell-Depleted Graft With Additional Infusion of Conventional T Cells and Regulatory T Cells, or Standard-of-Care Allogeneic Graft
Brief Title: Precision-T: A Study of Orca-T in Recipients Undergoing Allogeneic Transplantation for Hematologic Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Orca Biosystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Precision-T (PhIb component)
Record Dates: First submitted 2019-07-03; First posted 2019-07-10 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoid Leukemia; Myelodysplastic Syndromes; Acute Leukemia; Blastic Plasmacytoid Dendritic Cell Neoplasm (BPDCN); Chronic Myeloid Leukemia
Keywords: hematopoietic stem cell transplantation; acute leukemia; Myelodysplastic syndromes; matched related donor; matched unrelated donor
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Blastic Plasmacytoid Dendritic Cell Neoplasm; Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Subjects with Acute Leukemia or Myelodysplastic Syndrome, or BPDCN (Experimental): This is a non-randomized, single-arm study. All enrolled subjects will receive an allogeneic HCT with the Orca-T product.
  Interventions: Biological: Orca-T

INTERVENTIONS:
Biological: Orca-T — an allogeneic stem cell and T-cell immunotherapy biologic

SUMMARY:
This study will evaluate the safety, tolerability, and efficacy of Orca-T, an allogeneic stem cell and T-cell immunotherapy biologic manufactured for each patient (transplant recipient) from the mobilized peripheral blood of a specific, unique donor. It is composed of purified hematopoietic stem and progenitor cells (HSPCs), purified regulatory T cells (Tregs), and conventional T cells (Tcons) in participants undergoing myeloablative allogeneic hematopoietic cell transplant transplantation for hematologic malignancies.

ELIGIBILITY:
Key Inclusion Criteria:

Recipients must meet all of the following criteria:

1. Patients must diagnosed with one of the following histopathologically confirmed diseases, for which a myeloablative hematopoietic stem cell transplant (HCT) is planned:

   A) Acute myeloid, lymphoid, or mixed phenotype/undifferentiated leukemia who are not in CR or CRi (active disease) and/or MDS with >10% to <20% bone marrow blast burden (ages 18 to 75 years)

   B) Acute leukemia in CR/CRi or MDS that is DRI intermediate to high risk (ages 66 to 75 years)

   C) BPDCN (ages 18 to 65 years)

   D) Participants aged 18 to 65 who would be eligible for the Phase 3 component of Precision-T except for mild impairments of renal and/or hepatic function as defined by an eGFR of 50 to <60 mL/min and/or a total bilirubin of >ULN to ≤2 x ULN and diagnosed with either of the following:

   i. Acute myeloid, lymphoid, or mixed phenotype/undifferentiated leukemia that is in CR/CRi and DRI intermediate to high risk

   a) MDS that is DRI intermediate to high risk

   E) Acute or chronic leukemia in remission that is DRI low risk (ages 18 to 65 years), including the following:

   i. CML in chronic phase but with a history of accelerated phase or blast crisis or who are resistant to or intolerant of more than 1 first- and second-generation tyrosine kinase inhibitors

   ii. Acute myeloid leukemia (AML) with inv(16) without accompanying complex cytogenetics
2. Patients must be matched to a 8/8 HLA-matched related or unrelated donor
3. Estimated glomerular filtration rate (eGFR) > 50 mL/minute
4. Cardiac ejection fraction at rest ≥ 45% or shortening fraction of ≥ 27% by echocardiogram or radionuclide scan (MUGA)
5. Diffusing capacity of the lung for carbon monoxide (DLCO) (adjusted for hemoglobin) ≥ 50%
6. Total bilirubin < 2 times upper limit of normal (ULN) (patients with Gilbert's syndrome may be included where hemolysis has been excluded) and ALT/AST < 3 times ULN

Key Exclusion Criteria:

Recipients meeting any of the following exclusion criteria will not be eligible:

1. History of prior allogeneic HCT
2. Currently receiving corticosteroids or other immunosuppressive therapy. Topical corticosteroids or oral systemic corticosteroid doses less than or equal to 10 mg/day are allowed.
3. Pre-planned donor lymphocyte infusion (DLI)
4. Planned pharmaceutical in vivo or ex vivo T cell depletion
5. Positive for anti-donor HLA antibodies against an allele in the selected donor
6. Karnofsky performance score < 70%
7. Hematopoietic cell transplantation-specific Comorbidity Index (HCT-CI) > 4
8. Uncontrolled bacterial, viral or fungal infections (currently taking antimicrobial therapy and with progression or no clinical improvement) at time of enrollment
9. Seropositive for HIV-1 or -2 antibody, HTLV-1 or -2 antibody, Hepatitis B sAg, or Hepatitis C antibody
10. Any uncontrolled autoimmune disease requiring active immunosuppressive treatment
11. Concurrent malignancies or active disease within 1 year, except non-melanoma skin cancers that have been curatively resected
12. Women who are pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2019-11-21 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
The incidence of primary graft failure | 365 days
  The incidence of primary graft failure
The incidence of grade 3 or 4 aGVHD | 180 days
  The incidence of grade 3 or 4 aGVHD

SECONDARY OUTCOMES:
1-year overall survival (OS) | 365 days
  1-year overall survival (OS)
1 year graft-versus-host-disease-free and relapse-free survival (GRFS) | 365 days
  1 year graft-versus-host-disease-free and relapse-free survival (GRFS)
incidence and severity of acute and chronic graft vs host disease (GvHD) | 365 days
  incidence and severity of acute and chronic graft vs host disease (GvHD)
incidence of serious infections | 365 days
  incidence of serious infections
incidence of engraftment | 28 days
  incidence of engraftment of platelets and neutrophils

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - City of Hope, Duarte, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UC Davis, Sacramento, California
  - Stanford Health Care, Stanford, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - University of Miami Hospital and Clinics - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - The University of Kansas Hospital, Kansas City, Kansas
  - Massachusetts, Boston, Massachusetts
  - University of Michigan Health System - Michigan Medicine, Ann Arbor, Michigan
  - Weill Cornell Medicine - New York-Presbyterian Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Oregon Health & Sciences University - Knight Cancer Institute, Portland, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Utah - Huntsman Cancer Institute, Salt Lake City, Utah